CLINICAL TRIAL: NCT05428930
Title: A Randomized, Double-blind, Active-controlled, Single-center Phase I Trial to Investigate the Safety and Efficacy of CKDB-501B in Subjects With Moderate-to-severe Glabellar Lines
Brief Title: Safety and Efficacy of CKDB-501B in Subjects With Moderate-to-severe Glabellar Lines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CKD Bio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKDB-BAGL-102
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Glabellar Lines

STUDY DESIGN:
Intervention Model Description: Active-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKDB-501B (Experimental)
  Interventions: Drug: CKDB-501B
- Botox® 50U (Active Comparator)
  Interventions: Drug: Botox®50U

INTERVENTIONS:
Drug: CKDB-501B — Intramuscular injection CKDB-501B
  Arms: CKDB-501B
Drug: Botox®50U — Intramuscular injection Botox®50U
  Arms: Botox® 50U

SUMMARY:
A single-center, randomized, double-blind, single-injection, active-controlled, parallel-design study to evaluate the safety and efficacy of CKDB-501B in Glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with at least moderate glabellar frown lines at maximum frown using the severity score of at least 2(moderate) on the Facial Wrinkle Scale (4-point FWS)

Exclusion Criteria:

* Any medical condition (e.g., myasthenia gravis, Lambert-Easton syndrome, amyotrophic lateral sclerosis, etc.) that can affect the neuromuscular function
* History of facial nerve paralysis or ptosis
* Significant facial asymmetry
* Subjects with skin abnormalities such as infection, dermatologic disorders, scars, etc. at potential injection sites
* Previous treatment with any serotype of botulinum toxin products within 24 weeks (6 months) prior to Screening or planning to receive treatment with botulinum toxin during the study period
* Previous treatment with retinoids (isotretinoin, alitretinoin, etc.)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | [Time Frame: up to week 12]
  Severity and frequency of reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: beomjoon Kim, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No